CLINICAL TRIAL: NCT01208727
Title: The POSTCONDITIONING and THE NO REFLOW Phenomenon in Acute Myocardial Infarction
Brief Title: Post Cond No Reflow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-504
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Reperfusion Injury
Keywords: Myocardial infarction; Postconditioning; Microvascular obstruction; No reflow; MRI
MeSH Terms: conditions — Myocardial Reperfusion Injury; Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): 22 controls patients without post conditionment
- Intervention (Experimental): 22 posconditioned patients
  Interventions: Procedure: postconditioning

INTERVENTIONS:
Procedure: postconditioning — Direct postconditioning (brief repeated cycle of 4 occlusion and desocclusion of the initially occluded culprit coronary artery) after primary direct stenting.
  Arms: Intervention

SUMMARY:
After having shown that postconditioning allowed a significant 36% reduction of infarct size as assessed by blood levels of myocardial enzymes in acute myocardial patients, the investigators objective is to assess the effect of postconditioning in acute myocardial infarction (AMI) patients on microvascular obstruction lesions defined by cardiac MRI images.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old,
* Male or female,
* Presenting first myocardial infarction, with the beginning of pains < 12 hours,
* Requiring a revascularisation by primary angioplasty or " rescue " (after failure of thrombolysis) on IVA or RCA (not CA).
* Artery guilty with TIMI flow = 0

Exclusion Criteria:

* cardiac arrest before the angioplasty,
* Cardiogenic shock
* Occlusion of the artery circumflex responsible for the infarction
* Magnetic resonance imaging: contre indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Extent of the area of microvascular obstruction | 5 days
  Extent of the area of microvascular obstruction defined on post-gadolinium CMR images realized 48-72 hours after admission in each group

SECONDARY OUTCOMES:
Size of the myocardial infarction | 5 days
  Size of the myocardial infarction defined on post-gadolinium CMR images realized 48-72 hours after admission in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CROISILLE, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Thuny F, Lairez O, Roubille F, Mewton N, Rioufol G, Sportouch C, Sanchez I, Bergerot C, Thibault H, Cung TT, Finet G, Argaud L, Revel D, Derumeaux G, Bonnefoy-Cudraz E, Elbaz M, Piot C, Ovize M, Croisille P. Post-conditioning reduces infarct size and edema in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2012 Jun 12;59(24):2175-81. doi: 10.1016/j.jacc.2012.03.026. PMID 22676937